CLINICAL TRIAL: NCT01496430
Title: A Randomized, Double-Blind, Phase 3b Proof-of-Concept Study to Evaluate the Efficacy and Safety of TAK-491 Compared to Placebo When Used in Combination With Metformin in Subjects With Hypertension and Type 2 Diabetes
Brief Title: Efficacy and Safety of Azilsartan Medoxomil Used in Combination With Metformin in Participants With Hypertension and Diabetes
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business Decision; No Safety Or Efficacy Concerns. (See below)
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-491_304; U1111-1125-1197 (Registry Identifier: WHO)
Record Dates: First submitted 2011-12-18; First posted 2011-12-21 (Estimated); Results first posted 2015-05-06 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-04

CONDITIONS: Hypertension; Diabetes
Keywords: Drug Therapy; Hypertension and Diabetes
MeSH Terms: conditions — Hypertension; Diabetes Mellitus | interventions — azilsartan medoxomil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo QD (Placebo Comparator): Azilsartan medoxomil placebo-matching tablets, orally, once daily for up to 24 weeks.
  Interventions: Drug: Placebo
- Azilsartan Medoxomil 40 mg QD (Experimental): Azilsartan medoxomil 40 mg, tablets, orally, once daily for up to 24 weeks.
  Interventions: Drug: Azilsartan medoxomil
- Azilsartan Medoxomil 80 mg QD (Experimental): Azilsartan medoxomil 80 mg, tablets, orally, once daily for up to 24 weeks.
  Interventions: Drug: Azilsartan medoxomil

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo QD
Drug: Azilsartan medoxomil
  Other Names: TAK-491
  Arms: Azilsartan Medoxomil 40 mg QD
Drug: Azilsartan medoxomil
  Other Names: TAK-491
  Arms: Azilsartan Medoxomil 80 mg QD

SUMMARY:
The purpose of this study was to evaluate the antihypertensive and antiglycemic effects, as well as the safety and tolerability of TAK-491 (azilsartan medoxomil), once daily (QD), in stage 1 hypertensive, type 2 diabetes mellitus (T2DM) participants whose glycemic control was inadequate on metformin alone.

DETAILED DESCRIPTION:
The study included a Screening Period of up to 4 weeks, which coincided with a 2-week single-blind, placebo Run-in Period, a 24 week Treatment Period, and a 2-week Follow-up Period. The duration of the study was approximately 30 weeks. The planned number of participants (n=450) was not reached; actual enrollment consisted of 105 particpants. Due to low enrollment this study was terminated early by Takeda.

ELIGIBILITY:
Inclusion Criteria:

1. Was male or female and ≥18 years.
2. Had type 2 diabetes mellitus with HbA1c of ≥7.5 to ≤9.5% at Screening.
3. Was treated with metformin alone (no treatment with any antidiabetic agents other than metformin within the 3 months prior to Screening) and was experiencing inadequate glycemic control. The participant should have received metformin monotherapy for ≥8 weeks prior to Screening at a stable dose ≥1500 mg). Participants with a maximum tolerated dose (MTD) that was documented to be less than 1500 mg of metformin could also be enrolled if this dose had been stable for 8 weeks prior to Screening.
4. Was treated with antihypertensive therapy and had a mean, trough, sitting clinic systolic blood pressure (SBP) ≥135 and < 160 mm Hg on Day -1 (after washout of prior antihypertensive therapy) or the participant had not received antihypertensive treatment within 28 days before Screening and had a mean sitting clinic SBP ≥135 and < 160 mm Hg at the Screening Visit and on Day -1.
5. Had clinical laboratory evaluations (including clinical chemistry, hematology, and complete urinalysis) within the reference range for the testing laboratory or results that were deemed not clinically significant in this participant population for inclusion in this study, by the investigator.

Exclusion Criteria:

1. Had a mean, trough, sitting clinic diastolic blood pressure (DBP) ≥ 100 mm Hg at Day -1.
2. Had type 1 or poorly controlled type 2 diabetes mellitus (HbA1c >9.5%) at Screening.
3. Was taking or expected to take an excluded medication.
4. Had a history of myocardial infarction, heart failure, unstable angina, coronary artery bypass graft, percutaneous coronary intervention, hypertensive encephalopathy, cerebrovascular accident, or transient ischemic attack.
5. Had clinically significant cardiac conduction defects (for example, 3rd degree atrioventricular block, left bundle branch block, sick sinus syndrome, atrial fibrillation).
6. Had hemodynamically significant left ventricular outflow obstruction due to aortic valvular disease.
7. Had secondary hypertension of any etiology (e.g., renovascular disease, pheochromocytoma, Cushing's syndrome).
8. Had renal dysfunction defined as estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m2 at Screening.
9. Had albuminuria defined as >200 mg/g at Screening.
10. Had known or suspected unilateral or bilateral renal artery stenosis.
11. Had unexplained microhematuria ≥3 RBCs/HPF or macrohematuria at Screening and confirmed on repeat testing.
12. Treatment with antidiabetic agents (sulfonylureas, glucagon-like peptide-1 (GLP-1) analogues, dipeptidyl peptidase-4 (DPP-4) inhibitors, glinides, thiazolidinediones (TZDs), and/or insulin) other than metformin during the 3 months prior to Screening.
13. Had hyperkalemia as defined by central laboratory normal reference range at Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2012-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Director, Clinical Science, Study Director — Takeda
Locations (68):
- United States (68):
  - Birmingham, Alabama
  - Green Valley, Arizona
  - Tempe, Arizona
  - Tucson, Arizona
  - Buena Park, California
  - Hawaiian Gardens, California
  - Norwalk, California
  - Paramount, California
  - Rancho Cucamonga, California
  - Sacramento, California
  - San Diego, California
  - Tustin, California
  - Denver, Colorado
  - Bradenton, Florida
  - Brooksville, Florida
  - Hallandale, Florida
  - Jupiter, Florida
  - Miami, Florida
  - Orlando, Florida
  - Pembroke Pines, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Winter Park, Florida
  - Roswell, Georgia
  - Chicago, Illinois
  - Evergreen Park, Illinois
  - Gurnee, Illinois
  - Avon, Indiana
  - Greenfield, Indiana
  - Lexington, Kentucky
  - Paducah, Kentucky
  - Baltimore, Maryland
  - Columbia, Missouri
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Margate City, New Jersey
  - Albuquerque, New Mexico
  - Brooklyn, New York
  - Calabash, North Carolina
  - Greensboro, North Carolina
  - Lenoir, North Carolina
  - Morehead City, North Carolina
  - Salisbury, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Centerville, Ohio
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Downingtown, Pennsylvania
  - Fleetwood, Pennsylvania
  - Reading, Pennsylvania
  - Providence, Rhode Island
  - Anderson, South Carolina
  - Chattanooga, Tennessee
  - Kingsport, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Irving, Texas
  - North Richland Hills, Texas
  - Pearland, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Burke, Virginia
  - Manassas, Virginia
  - Richmond, Virginia
  - Virginia Beach, Virginia
  - Wauwatosa, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 41 investigative sites in the United States from 09 January 2012 to 30 May 2013.
Pre-assignment Details: Participants with a diagnosis of stage 1 essential hypertension and type 2 diabetes mellitus uncontrolled on metformin were enrolled equally in 1 of 3 treatment groups, once a day placebo, 40 mg or 80 mg TAK-491.
Period: Overall Study
Arm/Group | Placebo QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Started | 35 | 35 | 35
Completed | 29 | 30 | 25
Not Completed | 6 | 5 | 10
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Major Protocol Deviation | 0 | 0 | 1
Not completed — Lost to Follow-up | 2 | 3 | 1
Not completed — Voluntary Withdrawal | 2 | 1 | 6
Not completed — Principal Investigator Discretion | 0 | 1 | 1
Not completed — Other | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized Set includes all enrolled participants who were randomized via the Interactive Voice/Web Response System.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Total
Number analyzed (Participants) | 35 | 35 | 35 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (8.66) | 54.7 (7.63) | 55.8 (7.37) | 55.9 (7.89)
Age, Customized [Number; unit: participants]
  <45 years | 3 | 3 | 2 | 8
  Between 45 and 64 years | 25 | 29 | 30 | 84
  ≥65 years | 7 | 3 | 3 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 18 | 42
  Male | 21 | 25 | 17 | 63
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 11 | 15 | 14 | 40
  Non-Hispanic or Latino | 24 | 20 | 21 | 65
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 4 | 5 | 2 | 11
  Black or African American | 6 | 6 | 7 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  White | 25 | 23 | 26 | 74
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 35 | 105
Height [Mean (Standard Deviation); unit: cm] | 169.4 (9.81) | 169.8 (9.41) | 167.0 (12.30) | 168.8 (10.56)
Weight [Mean (Standard Deviation); unit: kg] | 93.41 (19.165) | 94.56 (20.084) | 92.33 (24.027) | 93.43 (21.012)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 32.50 (5.977) | 32.58 (5.475) | 32.94 (7.339) | 32.67 (6.255)
Smoking Classification [Number; unit: participants]
  Never smoked | 17 | 23 | 21 | 61
  Current smoker | 11 | 2 | 3 | 16
  Ex-smoker | 7 | 10 | 11 | 28
Baseline Glycosylated Hemoglobin (HbA1c) [Number; unit: participants]
  ≤8.5% | 24 | 24 | 20 | 68
  >8.5% | 11 | 11 | 15 | 37
Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: ml/min/1.73 m^2] | 87.86 (18.068) | 89.31 (15.631) | 89.72 (18.379) | 88.96 (17.253)
Estimated Glomerular Filtration Rate (eGFR) Categories [Number; unit: participants]
  30 - <60 mL/min/1.73 m^2 | 0 | 0 | 2 | 2
  60 - <90 mL/min/1.73 m^2 | 21 | 19 | 17 | 57
  ≥90 mL/min/1.73 m^2 | 14 | 16 | 16 | 46
Baseline Systolic Blood Pressure (SBP) Hypertension Severity Category [Number; unit: participants]
  SBP <140 mm Hg | 16 | 6 | 13 | 35
  140 ≤SBP <160 mm Hg | 19 | 23 | 16 | 58
  160 ≤SBP <180 mm Hg | 0 | 6 | 5 | 11
  SBP ≥ 180 mm Hg | 0 | 0 | 1 | 1
Baseline Diastolic Blood Pressure (DBP) Hypertension Severity Category [Number; unit: participants]
  DBP < 90 mm Hg | 25 | 18 | 25 | 68
  DBP ≥ 90 mm Hg | 10 | 17 | 10 | 37
Antihypertension Medication Within 28 Days [Number; unit: participants]
  Yes | 32 | 27 | 30 | 89
  No | 3 | 8 | 5 | 16
Washout Required [Number; unit: participants]
  21-Day Washout | 27 | 24 | 25 | 76
  4 Week Washout | 3 | 2 | 4 | 9
  Missing | 5 | 9 | 6 | 20
Female Reproductive Status [Number; unit: participants]
  Postmenopausal | 4 | 5 | 9 | 18
  Surgically Sterile | 6 | 3 | 8 | 17
  Female of Childbearing Potential | 4 | 2 | 1 | 7
  N/A (participant is male) | 21 | 25 | 17 | 63

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Sitting Clinic Systolic Blood Pressure
Description: The change in trough systolic blood pressure measured at week 8 relative to baseline. The trough is the average of the non-missing values of the 3 serial trough sitting systolic blood pressure measurements.
Time Frame: Baseline and Week 8
Population: The full analysis set included all randomized participants who took at least 1 dose of double-blind study medication. Missing values were imputed using last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 35 | 35 | 34
mm Hg | -3.1 (2.71) | -10.2 (2.69) | -13.6 (2.70)
Statistical Analysis 1: Comparison: Placebo QD vs Azilsartan Medoxomil 80 mg QD; Test type: Superiority or Other; p = 0.007, ANCOVA — Sequential testing was used to control for multiple comparisons. Azilsartan medoxomil 80 mg was first compared to placebo and if p-value ≤0.05 then azilsartaon medoxomil 40 mg was compared to placebo
Statistical Analysis 2: Comparison: Placebo QD vs Azilsartan Medoxomil 40 mg QD; Test type: Superiority or Other; p = 0.067, ANCOVA — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c)
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 24 relative to baseline.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage glycosylated hemoglobin
Arm/Group | Placebo QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 35 | 35 | 33
percentage glycosylated hemoglobin | 0.12 (0.174) | -0.19 (0.174) | 0.07 (0.179)
Statistical Analysis 1: Comparison: Placebo QD vs Azilsartan Medoxomil 80 mg QD; Test type: Superiority or Other; p = 0.860, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Azilsartan Medoxomil 40 mg QD; Test type: Superiority or Other; p = 0.210, ANCOVA — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in Trough Sitting Clinic Diastolic Blood Pressure
Description: The change in trough diastolic blood pressure measured at week 8 relative to baseline. The trough is the average of the non-missing values of the 3 serial trough sitting diastolic blood pressure measurements.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 35 | 35 | 34
mm Hg | -0.8 (1.36) | -5.4 (1.37) | -5.8 (1.37)

4. Secondary Outcome: Change From Baseline in the 24-hour Mean Systolic Blood Pressure, as Measured by Ambulatory Blood Pressure Monitoring
Description: The change in 24-hour mean systolic blood pressure measured at week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 24-hour mean is the average of all measurements recorded for 24 hours after dosing.
Time Frame: Baseline and Week 8
Population: The full analysis set included all randomized participants who took at least 1 dose of double-blind study medication. Observed cases.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 21 | 23 | 20
mm Hg | -1.6 (2.25) | -8.3 (2.15) | -11.3 (2.31)

5. Secondary Outcome: Change From Baseline in the 24-hour Mean Diastolic Blood Pressure, as Measured by Ambulatory Blood Pressure Monitoring
Description: The change in 24-hour mean diastolic blood pressure measured at week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 24-hour mean is the average of all measurements recorded for 24 hours after dosing.
Time Frame: Baseline and Week 8
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 21 | 23 | 20
mm Hg | -1.0 (1.28) | -4.7 (1.22) | -7.2 (1.31)

6. Secondary Outcome: Change From Baseline in the Mean Daytime (6 AM to 10 PM) Systolic Blood Pressure, as Measured by Ambulatory Blood Pressure Monitoring
Description: The change in daytime (6am to 10pm) mean systolic blood pressure measured week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Daytime mean is the average of all measurements recorded between the hours of 6 am and 10 pm.
Time Frame: Baseline and Week 8
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 21 | 23 | 20
mm Hg | -2.0 (2.23) | -9.0 (2.13) | -11.7 (2.28)

7. Secondary Outcome: Change From Baseline in the Mean Daytime (6 AM to 10 PM) Diastolic Blood Pressure, as Measured by Ambulatory Blood Pressure Monitoring
Description: The change in daytime (6am to 10pm) mean diastolic blood pressure measured at week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Daytime mean is the average of all measurements recorded between the hours of 6 am and 10 pm.
Time Frame: Baseline and Week 8
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 21 | 23 | 20
mm Hg | -1.4 (1.25) | -5.1 (1.20) | -7.5 (1.28)

8. Secondary Outcome: Change From Baseline in the Mean Nighttime (12 AM to 6 AM) Systolic Blood Pressure, as Measured by Ambulatory Blood Pressure Monitoring
Description: The change in nighttime (12am to 6am) mean systolic blood pressure measured at week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Nighttime mean is the average of all measurements recorded between the hours of 12 am and 6 am.
Time Frame: Baseline and Week 8
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 21 | 23 | 20
mm Hg | 0.4 (2.68) | -6.2 (2.57) | -10.9 (2.76)

9. Secondary Outcome: Change From Baseline in the Mean Nighttime (12 AM to 6 AM) Diastolic Blood Pressure, as Measured by Ambulatory Blood Pressure Monitoring
Description: The change in nighttime (12am to 6am) mean diastolic blood pressure measured at week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Nighttime mean is the average of all measurements recorded between the hours of 12 am and 6 am.
Time Frame: Baseline and Week 8
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 21 | 23 | 20
mm Hg | 0.6 (1.65) | -3.2 (1.58) | -7.2 (1.69)

10. Secondary Outcome: Change From Baseline in the 12-hr Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring
Description: The change in 12-hour mean systolic blood pressure measured at week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 12-hour mean is the average of all measurements recorded during the first 12 hours after dosing.
Time Frame: Baseline and Week 8
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 21 | 23 | 20
mm Hg | -2.7 (2.40) | -8.6 (2.29) | -12.3 (2.45)

11. Secondary Outcome: Change From Baseline in the 12-hr Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring
Description: as for outcome 10
Time Frame: Baseline and Week 8
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 21 | 23 | 20
mm Hg | -1.9 (1.37) | -4.7 (1.31) | -8.2 (1.40)

12. Secondary Outcome: Change From Baseline in the Trough (22 to 24 Hours After Dosing) Systolic Blood Pressure as Measured by Ambulatory Blood Pressure Monitoring
Description: The change in trough systolic blood pressure measured at week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The trough is the average of all measurements recorded from 22 to 24 hours after dosing.
Time Frame: Baseline and Week 8
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 21 | 23 | 20
mm Hg | 2.3 (2.80) | -7.6 (2.67) | -7.9 (2.87)

13. Secondary Outcome: Change From Baseline in the Trough (22 to 24 Hours After Dosing) Diastolic Blood Pressure as Measured by Ambulatory Blood Pressure Monitoring
Description: The change in trough diastolic blood pressure measured at week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The trough is the average of all measurements recorded from 22 to 24 hours after dosing.
Time Frame: Baseline and Week 8
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 21 | 23 | 20
mm Hg | 0.2 (1.63) | -6.8 (1.57) | -4.0 (1.66)

14. Secondary Outcome: Percentage of Participants Requiring Rescue Glycemic Therapy
Description: Percentage of participants requiring rescue glycemic therapy during study.
Time Frame: 24 Weeks
Population: The full analysis set included all randomized participants who took at least 1 dose of double-blind study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 35 | 35 | 35
percentage of participants | 25.7 | 25.7 | 25.7

15. Secondary Outcome: Time to First Glycemic Rescue
Description: The time to the first instance of participants requiring glycemic rescue during study.
Time Frame: 24 Weeks
Population: The full analysis set included all randomized participants who took at least 1 dose of double-blind study medication.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Placebo QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 35 | 35 | 35
Days | NA [21.57 to NA] — Median and third quartile times to glycemic rescue were not observed. | NA [22.57 to NA] — Median and third quartile times to glycemic rescue were not observed. | NA [17.14 to NA] — Median and third quartile times to glycemic rescue were not observed.

16. Secondary Outcome: Change From Baseline in HbA1c
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at each week indicated relative to baseline.
Time Frame: Baseline and Weeks 2, 4, 6, 8, 12, 16 and 20
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage glycosylated hemoglobin
Arm/Group | Placebo QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 35 | 35 | 33
percentage glycosylated hemoglobin
  Week 2 (n=34, 35, 32) | -0.01 (0.072) | 0.05 (0.071) | -0.06 (0.074)
  Week 4 (n=35, 35, 33) | -0.02 (0.093) | -0.02 (0.093) | 0.29 (0.096)
  Week 6 (n=35, 35, 33) | 0.06 (0.123) | -0.02 (0.123) | 0.24 (0.127)
  Week 8 (n=35, 35, 33) | 0.05 (0.137) | -0.03 (0.138) | 0.23 (0.141)
  Week 12 (n=35, 35, 33) | 0.00 (0.171) | -0.05 (0.171) | 0.29 (0.176)
  Week 16 (n=35, 35, 33) | 0.09 (0.171) | -0.06 (0.171) | 0.16 (0.176)
  Week 20 (n=35, 35, 33) | 0.14 (0.167) | -0.13 (0.168) | 0.09 (0.172)

17. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose
Description: The change between the fasting plasma glucose value collected at each week indicated relative to baseline.
Time Frame: Baseline and Weeks 2, 4, 6, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 35 | 35 | 34
mmol/L
  Week 2 (n=34, 35, 34) | 0.16 (0.435) | 0.64 (0.429) | 1.03 (0.435)
  Week 4 (n=35, 35, 34) | 0.96 (0.464) | 0.45 (0.464) | 0.81 (0.470)
  Week 6 (n=35, 35, 34) | 0.71 (0.445) | 0.28 (0.445) | 0.81 (0.451)
  Week 8 (n=35, 35, 34) | 0.39 (0.368) | 0.34 (0.368) | 0.96 (0.373)
  Week 12 (n=35, 35, 34) | 0.76 (0.417) | 0.09 (0.417) | 0.94 (0.423)
  Week 16 (n=35, 35, 34) | 0.36 (0.379) | 0.17 (0.379) | 0.49 (0.384)
  Week 20 (n=35, 35, 34) | 0.94 (0.438) | 0.01 (0.438) | 0.86 (0.444)
  Week 24 (n=35, 35, 34) | 0.76 (0.459) | -0.15 (0.459) | 0.48 (0.465)

18. Secondary Outcome: Change From Baseline to Week 6 and Week 24 in 2h Glucose During Oral Glucose Tolerance Testing (OGTT)
Description: The change between the glucose value collected at weeks 6 and 24 relative to baseline. Oral glucose tolerance test measures glucose, insulin, C-peptide, insulin/glucose ratio, and glucagon through blood samples drawn at 0, 30, 60, and 120 minutes following consumption of a 75 g glucose beverage.
Time Frame: Baseline and Weeks 6 and 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 32 | 31 | 29
mmol/L
  Week 6 (n=30, 30, 29) | 1.01 (0.555) | -0.46 (0.556) | -0.09 (0.565)
  Week 24 (n=25, 26, 19) | -0.44 (0.824) | -1.66 (0.811) | -3.94 (0.949)

19. Secondary Outcome: Change From Baseline to Week 6 and Week 24 in the Area Under the Plasma Concentration-time Curve (AUC) for Glucose During OGTT
Description: The change between the AUC for glucose at weeks 6 and 24 relative to baseline. AUC will be calculated based on measurements at 0, 30, 60 and 120 minutes. Oral glucose tolerance test measures glucose, insulin, C-peptide, insulin/glucose ratio, and glucagon through blood samples drawn at 0, 30, 60, and 120 minutes following consumption of a 75 g glucose beverage.
Time Frame: Baseline and Weeks 6 and 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mmol*hours/L
Arm/Group | Placebo QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 30 | 31 | 29
mmol*hours/L
  Week 6 (n=28, 29, 29) | 1.60 (1.159) | -1.01 (1.148) | 1.04 (1.140)
  Week 24 (n=23, 24, 19) | -1.97 (1.339) | -1.13 (1.308) | -5.52 (1.471)

20. Secondary Outcome: Change From Baseline to Week 6 and Week 24 in AUC for Insulin During OGTT
Description: The change between the AUC for insulin at weeks 6 and 24 relative to baseline. AUC will be calculated based on measurements at 0, 30, 60 and 120 minutes. Oral glucose tolerance test measures glucose, insulin, C-peptide, insulin/glucose ratio, and glucagon through blood samples drawn at 0, 30, 60, and 120 minutes following consumption of a 75 g glucose beverage.
Time Frame: Baseline and Weeks 6 and 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: pmol*hours/L
Arm/Group | Placebo QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 29 | 32 | 28
pmol*hours/L
  Week 6 (n=28, 31, 28) | 64.4 (74.80) | -26.1 (71.42) | 19.5 (74.78)
  Week 24 (n=21, 25, 19) | -63.3 (162.81) | 80.1 (149.88) | 477.0 (169.22)

21. Secondary Outcome: Change From Baseline to Week 6 and Week 24 in AUC for C-peptide During OGTT
Description: The change between the AUC for C-peptide at weeks 6 and 24 relative to baseline. AUC will be calculated based on measurements at 0, 30, 60 and 120 minutes. Oral glucose tolerance test measures glucose, insulin, C-peptide, insulin/glucose ratio, and glucagon through blood samples drawn at 0, 30, 60, and 120 minutes following consumption of a 75 g glucose beverage.
Time Frame: Baseline and Weeks 6 and 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: nmol*hours/L
Arm/Group | Placebo QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 29 | 32 | 28
nmol*hours/L
  Week 6 (n=28, 31, 28) | 0.051 (0.1779) | -0.091 (0.1696) | -0.138 (0.1780)
  Week 24 (n=21, 25, 19) | -0.449 (0.2323) | 0.182 (0.2138) | 0.155 (0.2444)

22. Secondary Outcome: Change From Baseline to Week 6 and Week 24 in AUC for Insulin/Glucose Ratio During OGTT
Description: The change between the AUC for insulin/glucose ratio at weeks 6 and 24 relative to baseline. AUC will be calculated based on measurements at 0, 30, 60 and 120 minutes. Oral glucose tolerance test measures glucose, insulin, C-peptide, insulin/glucose ratio, and glucagon through blood samples drawn at 0, 30, 60, and 120 minutes following consumption of a 75 g glucose beverage.
Time Frame: Baseline and Weeks 6 and 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: pmol*hr/mmol
Arm/Group | Placebo QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 28 | 31 | 28
pmol*hr/mmol
  Week 6 (n=27, 29, 28) | 4.86 (5.777) | 1.73 (5.578) | -0.75 (5.663)
  Week 24 (n=20, 23, 19) | -5.36 (14.823) | 1.05 (13.883) | 52.68 (14.976)

23. Secondary Outcome: Change From Baseline to Week 6 and Week 24 in AUC for Glucagon During OGTT
Description: The change between the AUC for glucagon at weeks 6 and 24 relative to baseline. AUC will be calculated based on measurements at 0, 30, 60 and 120 minutes. Oral glucose tolerance test measures glucose, insulin, C-peptide, insulin/glucose ratio, and glucagon through blood samples drawn at 0, 30, 60, and 120 minutes following consumption of a 75 g glucose beverage.
Time Frame: Baseline and Weeks 6 and 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: ng*hours/L
Arm/Group | Placebo QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 30 | 30 | 28
ng*hours/L
  Week 6 (n=27, 27, 27) | -5.8 (9.34) | 27.1 (9.39) | 0.2 (9.32)
  Week 24 (n=22, 23, 19) | 2.7 (8.51) | 12.0 (8.45) | 1.0 (9.34)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 14 days (or 30 days for a serious adverse event) after the last dose of double-blind study drug, for up to 28 weeks.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Serious Adverse Events (participants affected / at risk) | 0/35 | 1/35 | 0/35
Other Adverse Events (participants affected / at risk) | 10/35 | 10/35 | 8/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo QD (N=35) | Azilsartan Medoxomil 40 mg QD (N=35) | Azilsartan Medoxomil 80 mg QD (N=35)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo QD (N=35) | Azilsartan Medoxomil 40 mg QD (N=35) | Azilsartan Medoxomil 80 mg QD (N=35)
Urinary tract infection (Infections and infestations) | 3 | 4 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 2
Constipation (Gastrointestinal disorders) | 2 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Proteinuria (Renal and urinary disorders) | 2 | 0 | 0

LIMITATIONS AND CAVEATS:
Because of low enrollment in the study, the sample sizes in the results data do not allow for significant interpretation of the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.